CLINICAL TRIAL: NCT01725854
Title: Relaxation Response (RR) Training for PTSD Prevention in Soldiers a.k.a. "SPIRIT SMART" (Stemming PTSD, Increasing Resilience and Impeding Trauma in Service Members: Assessing Relaxation Response Training)
Brief Title: Relaxation Response Training for PTSD Prevention in US Military Personnel
Acronym: RR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of staff for completion
Sponsor: William Beaumont Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: W81XWH-10-1-1011/ 367294
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Relaxation Response Training (Experimental): The Military tailored RR training program will consist of six weekly small group sessions which involve group presentations, in-group skill building exercises, and at-home assignments. Groups will contain 5-8 participants who are active-duty Soldiers enrolled in either Respect-MIL or the Interdisciplinary Pain Management Center (IPMC).
  Interventions: Behavioral: Relaxation Response training
- Standard of Care (No Intervention): Participants randomized to the control group will receive standard care through their providers at Respect-MIL or at the IPMC. Participants randomized to the control group will remain on the wait list for further standard care. After the collection of the final data point, these participants will also have the option to participate in an abbreviated, two-hour version of the RR training.

INTERVENTIONS:
Behavioral: Relaxation Response training — Behavioral Relaxation Response Training (Benson-Henry Institute Relaxation Response Training) Participants randomized to the intervention group will participate in the six weekly RR sessions. Examples of in-group skill building exercises are mini relaxations, diaphragmatic breathing, introduction to imagery, and eliciting RR through Yoga. Presentations topics include Introduction to Mind/Body Medicine, Introduction to the RR, Experiential RR Sessions, and Introduction to Cognitive Restructuring. Home skill building assignments include relaxation focus practice, an appreciation journal, self-monitoring with Biodots (biosensor technology that helps participants to monitor and regulate their psycho-emotional state), physical activity, balanced nutrition, and progress notes.
  Other Names: Benson-Henry Institute Relaxation response training
  Arms: Relaxation Response Training

SUMMARY:
The purposes of this study are to evaluate the acceptability and utility of a mind-body intervention on a convenience sample of Soldiers (n=120) who have screened positive through RESPECT-MIL for symptoms that may lead to post-traumatic stress and to test the effectiveness of this Relaxation Response (RR) intervention designed to decrease the physiological and psychosocial effects of stress and trauma. The study aims to enhance the psychological health of Soldiers with a RR intervention designed to promote self-awareness of physiological responses to stress and the ability to increase relaxation responses.

DETAILED DESCRIPTION:
Specific Aims:

1. Demonstrate that trainers can be trained effectively to deliver the intervention, a mind-body skills training program based on the Benson-Henry Institute's standard RR training curriculum and tailored to a military population.
2. Evaluate feasibility, acceptability, and compliance to the training program in an active duty military population.
3. Compare outcomes on sleep disturbance, PTSD, stress-related symptoms, quality of life, and psychosocial variables related to resilience of Soldiers who receive the 6-week training program to promote the Relaxation Response to those Soldiers who do not receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, male and female volunteer individual military Service Members, DoD civilians or approved contractors working for DoD, primarily from multidisciplinary healthcare providers.
* Willingness to participate in the research project.
* Committed to the entire period of time of the research project.
* Currently working or stationed at Ft Bliss, Texas.
* No impending orders for deployment/ TDY/ PCS/ ETS or retirement for at least 8 weeks from the day of study enrollment.
* Able to read and speak English.
* Capable to consent.

Exclusion Criteria:

• Diagnosed with severe PTSD or other mental health issues disclosed as self-reported

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Sleep | 6 weeks
  Sleep will be measured pre and post intervention. Sleep will be measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI assesses sleep quality and disturbances during the past month based on seven component scores for sleep quality, latency, duration, efficiency, disturbance, medication use, and daytime dysfunction that sum to a global score. A Sleep Diary will also be used to measure sleep and related factors.

SECONDARY OUTCOMES:
Anger | 6 Weeks
  Anger, measured with the Spielberger State-Trait Anger Expression Inventory-2 (STAXI-2)
Health Status | 6 Weeks
  Health Status as measured with the Veterans RAND 12-item Health Survey Short Form (VR-12 or SF-12) and the Functional Assessment of Chronic Illness Therapy- Spiritual Well-Being 12 (Non-Illness)
Resilience | 6 Weeks
  Resilience will be measured with the Post Traumatic Growth Inventory
Stress | 6 Weeks
  Stress as measured with physiological measurements of blood pressure and heart rate (pulse) and subjective measurement using the Perceived Stress Scale

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Petri, MD, Principal Investigator — William Beaumont Army Medical Center
Locations (1):
- William Beaumont Army Medical Center, Ft Bliss, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study terminated